CLINICAL TRIAL: NCT01688609
Title: Phase II Study of Lapatinib and Trastuzumab Followed by Concurrent Lapatinib, Trastuzumab, and Paclitaxel Followed by Surgery for Primary HER2-positive (HER2+) Breast Cancer
Brief Title: Lapatinib Ditosylate, Trastuzumab, Paclitaxel, and Surgery in Treating Patients With Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01970; NCI-2012-01970 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000734375; ACE-001 (Other: Saint Luke's International Hospital); 9020 (Other: CTEP)
Record Dates: First submitted 2012-09-16; First posted 2012-09-20 (Estimated); Results first posted 2017-09-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-08

CONDITIONS: HER2-positive Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib; N-(3-chloro-4-((3-fluorobenzyl)oxy)phenyl-6-(5-((methylsulfonyl)ethyl)aminomethyl)-2-furyl)-4-quinazolinamine; Paclitaxel; Taxes; Trastuzumab

ARMS (1):
- Treatment (lapatinib, trastuzumab, paclitaxel, surgery) (Experimental): Drug exposure: Patients receive lapatinib ditosylate PO QD and trastuzumab IV over 30-90 minutes once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Preoperative therapy: Patients receive lapatinib ditosylate PO QD, trastuzumab IV over 30 minutes once weekly, and paclitaxel IV over 90 minutes once weekly for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo lumpectomy or mastectomy.
  Interventions: Drug: lapatinib ditosylate; Drug: paclitaxel; Biological: trastuzumab; Procedure: therapeutic conventional surgery; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lapatinib ditosylate — Given PO
  Other Names: GSK572016; GW-572016; GW2016; Lapatinib; Tykerb
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Procedure: therapeutic conventional surgery — Undergo lumpectomy or mastectomy
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving lapatinib ditosylate together with trastuzumab, paclitaxel, and surgery works in treating patients with breast cancer. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as trastuzumab, can block tumor growth in different ways. Some block the ability of tumor to grow and spread. Others find tumor cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the changes in cancer stem cell (CSC) markers; % CD44 variant (CD44v)-positive tumor cells and aldehyde dehydrogenase-1 (ALDH1) positivity before and after study drug exposure and after concurrent preoperative chemotherapy.

II. To determine the pathological complete response (pCR) rate produced by lapatinib (lapatinib ditosylate) + trastuzumab followed by concurrent preoperative lapatinib, trastuzumab, and paclitaxel chemotherapy for operable human epidermal growth factor receptor 2-positive (HER2+) breast cancer.

SECONDARY OBJECTIVES:

I. To determine the cellular response rate produced by study drug exposure and/or concurrent preoperative chemotherapy.

II. To determine cutoff values of baseline ratios of phosphorylated HER2 (pHER2)/HER2, phosphorylated epidermal growth factor receptor (EGFR) (pEGFR)/EGFR, phosphorylated ERK (pERK)/ERK and phosphorylated protein kinase B (pAkt)/Akt that are associated with pCR.

III. To assess the safety and tolerability of study therapy in Japanese women.

OUTLINE:

Drug exposure: Patients receive lapatinib ditosylate orally (PO) once daily (QD) and trastuzumab intravenously (IV) over 30-90 minutes once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.

Preoperative therapy: Patients receive lapatinib ditosylate PO QD, trastuzumab IV over 30 minutes once weekly, and paclitaxel IV over 90 minutes once weekly for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo lumpectomy* or mastectomy*.

After completion of study treatment, patients are followed up for 12 weeks.

NOTE: * Patients considered to be candidates for breast-conservation therapy (BCT) are offered lumpectomy. Patients who are not considered to be candidates for BCT or who do not desire BCT undergo total mastectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed primary invasive breast cancer
* Primary tumor is larger than 2 cm in diameter (T2) as measured by caliper or ultrasound
* Overexpression and/or amplification of HER2 is confirmed by immunohistochemistry (IHC) 3+ or fluorescence in situ hybridization (FISH) + when IHC 2+
* Patients have not received prior therapies for breast cancer
* Patients have Karnofsky >= 70%
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9.0 g/dL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 times institutional upper limit of normal
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvate transaminase[SGPT]) =< 2.5 times institutional ULN
* Creatinine =< 1.5 times institutional upper limit of normal (ULN)
* Patients must have left ventricular ejection fraction (LVEF) >= 50% by multi-gated acquisition (MUGA) or echocardiography
* Patients must be able to take oral medications (i.e., no uncontrolled vomiting, inability to swallow, or diagnosis of chronic malabsorption)
* Women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation as well as for at least 6 months after the last dose of trastuzumab
* Ability to understand and willingness not only for treatment but also for undergoing serial biopsies and sign a written informed consent document
* Only Japanese women are eligible for the trial

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy
* Patients who are receiving any other investigational agents
* Patients have distal metastasis (stage IV disease)
* Patients with previous (within 10 years) or current history of malignant neoplasm except for curatively treated basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to lapatinib or other agents used in study
* Patients receiving any medications or substances that are inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) are ineligible
* Patients who have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women
* Patients who have family or personal history of congenital long or short QT syndrome, Brugada syndrome, QT/QTc prolongation, or torsade de pointes
* Patients who have chronic gastrointestinal disease presenting with diarrhea (inflammatory bowel disease, malabsorption, or >= grade 2 diarrhea of any etiology at baseline)
* Patients who have neuropathy >= grade 2 of any cause
* Patients are diagnosed with inflammatory breast cancer or bilateral breast cancer

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2016-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teruo Yamauchi, Principal Investigator — Saint Luke's International Hospital
Locations (3):
- M D Anderson Cancer Center, Houston, Texas, United States
- Japan (2):
  - Keio University, Shinjuku-ku, Tokyo
  - Saint Luke's International Hospital, Chūōku, Toyko

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery): Drug exposure: Patients receive lapatinib ditosylate PO QD and trastuzumab IV over 30-90 minutes once weekly for 6 weeks in the absence of disease progression or unacceptable toxicity.
  Preoperative therapy: Patients receive lapatinib ditosylate PO QD, trastuzumab IV over 30 minutes once weekly, and paclitaxel IV over 90 minutes once weekly for 12 weeks in the absence of disease progression or unacceptable toxicity. Patients then undergo lumpectomy or mastectomy.
  lapatinib ditosylate: Given PO
  paclitaxel: Given IV
  trastuzumab: Given IV
  therapeutic conventional surgery: Undergo lumpectomy or mastectomy
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  Japan | 18

OUTCOME MEASURES:

1. Primary Outcome: Expression of ALDH1 and CD44v Change in the Binary Biomarkers From Baseline to 6 Weeks and 18 Weeks
Description: For biomarkers ALDH1 and CD44v, the change in the proportions of CD44v-positive (CD44v+) tumor cells and ALDH1-positive (ALDH1+) tumor cells in tumor tissue from baseline to 6 weeks and 18 weeks time points were determined for each patient. For biomarker change, changes in the binary biomarkers between time points were assessed using McNemar's test in all patients and separately in patients with and without pCR.
Time Frame: From baseline to 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
Number analyzed (Participants) | 18
Participants
  baseline CD44v expression : pCR | 5
  baseline CD44v expression : non-pCR | 3
  CD44v expression at 6 weeks : pCR | 0
  CD44v expression at 6 weeks : non-pCR | 4
  CD44v expression at 18 weeks : pCR | 0
  CD44v expression at 18 weeks : non-pCR | 5
  baseline ALDH1 expression : pCR | 8
  baseline ALDH1 expression : non-pCR | 10
  ALDH1 expression at 6 weeks : pCR | 7
  ALDH1 expression at 6 weeks : non-pCR | 10
  ALDH1 expression at 18 weeks : pCR | 8
  ALDH1 expression at 18 weeks : non-pCR | 9

2. Primary Outcome: Number of Participants With Pathological Complete Response (pCR)
Description: The point estimate of the pCR rate will be calculated for all patients. pCR is defined as the abscence of invasive cancer in the breast and regional lymph nodes following neoadjuvant chemotherapy.
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
Number analyzed (Participants) | 18
Participants | 8

3. Secondary Outcome: Cellular Response Rate, Defined as Patients With an Epithelial Phenotype Having Eradication of CTCs; Patients With a Mesenchymal Phenotype Having Eradication of Tumor Cells; Patients With a Mesenchymal Phenotype Converting to an Epithelial Phenotype
Description: Cellular response will be documented and calculated for rate in all patients.
Time Frame: Up to 18 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
Number analyzed (Participants) | 18
participants
  positive cellular response at 6 weeks | 4
  positive cellular response at 18 weeks | 10

4. Secondary Outcome: EGFR-mutation Status of Tumors and Changes in the Ratio of Phosphorylated to Nonphosphorylated HER2, EGFR, ERK, Akt, and the Ki67 and TUNEL Indices Before and After Treatment
Description: The EGFR mutation status will be a binary variable (yes vs. no), and the phosphorylation status of HER2 and EGFR will be a ratio variable (0-100%). The CART method to identify cut-off points for the phosphorylation ratio of molecules of interest will be used, such that ratios above the cut-off point will be considered "high phosphorylation" and ratios below the cut-off point will be considered "low phosphorylation."
Time Frame: From baseline to 24 weeks
Population: The study was not able to determine the cut off value of total and phorylated RTK ratio. Assays were not reliable. Data of EGFR mutations were not collected.
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of Participants With Treatment-Related Toxicities
Time Frame: Up to 12 weeks after completion of study treatment
Measure: Number; unit: participants
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
Number analyzed (Participants) | 18
participants
  Grade 3 ALT increase | 2
  Grade 3 GGT increase | 1
  Grade 3 leukopenia | 1
  Grade 3 neutropenia | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery)
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 17/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Lapatinib, Trastuzumab, Paclitaxel, Surgery) (N=18)
diarrhea (Gastrointestinal disorders) | 17
oral mucositis (Gastrointestinal disorders) | 14
hand-foot syndrome (Skin and subcutaneous tissue disorders) | 13
increased alanine aminotransferase level (Investigations) | 12
increased aspartate aminotransferase (Investigations) | 11
rash (Skin and subcutaneous tissue disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less